CLINICAL TRIAL: NCT03417297
Title: A Pilot Open-label Clinical Trial Evaluating the ExAblate Model 4000 Type-1 Focused Ultrasound Thalamotomy for the Prevention of Secondary Generalization in Focal Onset Epilepsy
Brief Title: A Pilot Study: Focused Ultrasound Thalamotomy for the Prevention of Secondary Generalization in Focal Onset Epilepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0350
Record Dates: First submitted 2018-01-10; First posted 2018-01-31 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Partial Seizures With Secondary Generalization; Focal Epilepsy With Secondary Generalization

STUDY DESIGN:
Intervention Model Description: This is a pilot study. Ten (10) adults with refractory, focal epilepsy with secondary generalization and able to provide informed consent will undergo focused ultrasound (FUS) thalamotomy. Initially, 3 participants will be enrolled and followed for 3 months to assess the safety of study intervention. Pending review by the Data and Safety Monitoring Committee (DSMC) and the US Food and Drug Administration (FDA), additional subjects will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- high intensity focused ultrasound (Experimental): Initially, 3 patients will be enrolled and followed for 3 months to assess the safety of study intervention which is unilateral focused ultrasound thalamotomy (anterior nucleus). These data will be reviewed by the Data and Safety Monitoring Committee (DSMC) and the FDA. If approval is granted by the DSMC and FDA, then additional subjects will be enrolled.
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — Participants will undergo high intensity focused ultrasound surgery utilizing magnetic resonance (MR) imaging guidance using a 3 Tesla scanner.
  Other Names: ExAblate Model 4000 Type-1 Focused Ultrasound

SUMMARY:
The purpose of this study is to assess the safety and feasibility of unilateral focused ultrasound thalamotomy in adults with focal onset epilepsy whose medicines are not working well. The ExAblate (ExAblate) transcranial system is the name of the device that will be used to create and send ultrasound waves through the scalp and skull precisely to a small structure located in the center of the brain. This structure is known as the "Anterior Nucleus", and is an important region in the brain that may cause seizures. Safety will be measured by recording and analyzing the frequency of side effects throughout participation. Feasibility will be measured by the ability to create a lesion in the anterior nucleus.

DETAILED DESCRIPTION:
This is an open-label prospective intervention study. Ten (10) adults with refractory, focal epilepsy with secondary generalization and able to provide informed consent will undergo focused ultrasound (FUS) thalamotomy. In addition to the diagnosis of medically refractory epilepsy, these patients will need to meet protocol specific inclusion and exclusion criteria. These adults will be screened from the patients being cared for by the epilepsy program at the University of North Carolina at Chapel Hill or referred from elsewhere for enrollment in the study. Initially, 3 participants will be enrolled and followed for 3 months to assess the safety of study intervention. Pending review by the Data and Safety Monitoring Committee (DSMC) and the US Food and Drug Administration (FDA), additional subjects will be enrolled.

This pilot study is being conducted to test the feasibility of this device in order to confirm the design and operating specifications of the device including the ability to identify and accurately ablate the target focus within the Anterior Nucleus.

Safety will be assessed by the frequency of side effects, e.g., new onset of neurological deficits, performance deterioration on neuropsychological testing. Feasibility is defined as the ability to create the desired lesion within the anterior nucleus.

Seizure frequency data will be collected by seizure questionnaire. Quality of life will be measured by the Quality of Life in Epilepsy Inventory (QOLIE-31). Imaging analysis will include a comparison of pre- and post-intervention imaging to identify brain networks associated with clinical outcomes and determine changes in resting-state functional connectivity (assessed by fMRI), as well as in structural (assessed by volumetric T1 and T2 weighted imaging) and microstructural (assessed by diffusion tensor imaging) brain anatomy.

Subject satisfaction with FUS thalamotomy will be assessed by the Epilepsy Surgery Satisfaction Questionnaire (ESSQ-19).

ELIGIBILITY:
Inclusion Criteria:

* Medically refractory epilepsy (≥2 antiepileptic drug failures) deemed disabling by the patient and study investigators.
* Focal seizures with secondary generalization; with or without primary generalized seizures.
* ≥ 3 seizures/month on average based on seizure diary of patient's preferred format during the three months prior to enrollment.
* Stable prescribed epilepsy medication dosages, including stopping or starting medication, for 3 months before enrollment.
* Anterior Nucleus (AN) identifiable on MRI (structural T1 and T2 images).
* Willing to maintain seizure diary (3 months before & 3 months after the study treatment).
* Involved caregiver such as a spouse, family member, or family friend willing to provide reliable care during the study participation.
* Ability to provide written informed consent to participate.
* Previous seizure work-up to include:

  1. Home EEG, Epilepsy Monitoring Unit (EMU) video EEG, or intracranial EEG.
  2. Baseline neuropsychological assessment, which includes the Wechsler Advanced Clinical Solutions - Test of Premorbid Functioning (TOPF). Participants obtaining an Intelligence Quotient (IQ) score of ≥70 on the TOPF will be included.
  3. High-definition MRI imaging/Position emission tomography (PET) imaging.

Exclusion Criteria:

* Have on average less than 3 seizures a month.
* Have an indwelling vagal nerve stimulator.
* Have severe untreated neuropsychiatric disorders (e.g., untreated depression or behavioral problems).
* History of drug or alcohol abuse in the last 12 months.
* Presence of primary generalized epilepsy (e.g., Lennox Gastaut, drop attacks).
* Presence of post-infectious epilepsy (i.e., epilepsy from post-herpetic encephalitis).
* Previous corpus callosotomy (surgery to cut the fibers, called the corpus callosum, that separate each half of the brain).
* Significant structural brain abnormalities.
* Unable or unwilling to maintain your current anti-seizure drug dosage for 3 months post-treatment.
* Pregnant or not practicing birth control methods.
* History of claustrophobia (fear of closed spaces).
* Presence of an MRI contraindicated implanted metal or medical device (e.g., pacemaker, metallic joints, or insulin pump).
* Uncontrolled hypertension or other comorbid conditions (e.g., uncontrolled heart or lung disease).
* Skull Density Ratio (SDR) <0.4.
* IQ score of <70 on the Wechsler Advanced Clinical Solutions - Test of Premorbid Functioning (TOPF), a measure conducted as part of baseline neuropsychological assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Successful Lesion Creation | during the surgical procedure
  Feasibility is defined as the ability to create the desired lesion within the anterior nucleus in 80% or more of participants.
Number of Participants with Adverse Events | 12 months
  Safety will be assessed by the frequency of side effects, e.g. new onset of neurological deficits, performance deterioration on neuropsychological testing.

SECONDARY OUTCOMES:
Change in Number of Seizures Reported Across Time | up to 24 months
  Captured by participant-recorded seizure questionnaires. Assessed at Baseline, Day 7, Day 30, and months 3, 6, 12 and 24.
Total QOLIE-31-P Score Across Time | up to 12 months
  The Quality of Life in Epilepsy Inventory-31-Problems (QOLIE-31-P) is a survey of health-related quality of life for adults with epilepsy. The QOLIE-31-P is completed by the patient. It contains 39 items, of which a total of 30 are used to make up 7 different subscales. Scores range from 0-100, with higher scores indicating a greater level of functioning and QoL. Assessed at Baseline, and months 1, 3, 6, and 12.
Change MRI parameter (water diffusivity) | Baseline, (Day 1), Month 3
  Water Diffusivity assessed by structural and microstructural MRI in a voxel-wise manner and compared between pre and post operative MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Vibhor Krishna, MD, SM, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krishna V, Mindel J, Sammartino F, Block C, Dwivedi AK, Van Gompel JJ, Fountain N, Fisher R. A phase 1 open-label trial evaluating focused ultrasound unilateral anterior thalamotomy for focal onset epilepsy. Epilepsia. 2023 Apr;64(4):831-842. doi: 10.1111/epi.17535. Epub 2023 Mar 1. PMID 36745000